CLINICAL TRIAL: NCT06406348
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 1, Single Ascending Dose Trial to Assess the Safety, Tolerability and Pharmacokinetic Effects of ALIA-1758 in Healthy Participants
Brief Title: A Phase 1 Trial to Assess Safety, Tolerability and Pharmacokinetics of ALIA-1758 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALIA-1758-101
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Single Ascending Dose (SAD) cohorts
  Interventions: Drug: ALIA-1758
- Placebo (Placebo Comparator): Single Ascending Dose (SAD) cohorts
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ALIA-1758 — Intravenous or subcutaneous doses
  Arms: Active
Other: Placebo — Intravenous or subcutaneous doses
  Arms: Placebo

SUMMARY:
This is a Phase 1, first in human (FIH), double-blind, placebo-controlled, single ascending dose (SAD) trial to assess the safety, tolerability, and pharmacokinetics (PK) of intravenously (IV) or subcutaneously (SC) injected ALIA-1758 in healthy male and female participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must understand the nature of the trial and must provide signed and dated written informed consent in accordance with local regulations before the conduct of any trial-related procedures.
* Healthy as determined by the Investigator, based on a medical evaluation including medical history, physical examination, laboratory tests and electrocardiogram (ECG) recording. A participant with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if, in the opinion of the Investigator, the finding is (a) unlikely to introduce additional risk to the participant, (b) will not interfere with trial procedures or confound trial results, and (c) is not otherwise exclusionary (see Exclusion Criteria).
* Body weight of at least 50.0 kg for men and 45.0 kg for women and Body Mass Index (BMI) within the range of 17.5-32.0 kg/m2 (inclusive) at Screening.

Key Exclusion Criteria:

* A history or presence of a clinically significant hepatic, biliary, renal, gastrointestinal, cardiovascular, endocrine, pulmonary, ophthalmologic, immunologic, hematologic, dermatologic, psychiatric, neurologic abnormality, or chronic urinary tract infections.
* A clinically significant abnormality on physical examination, ECG, or laboratory evaluations at Screening or between Screening and (first) dose administration.
* The participant is, in the opinion of the Investigator or Medical Monitor, unlikely to comply with the protocol or is unsuitable for any reason.

Other criteria may apply

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 85 days after dosing
  Incidence, severity, seriousness, and causality of treatment-emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Pharmacokinetic parameters of ALIA-1758 in healthy subjects: Cmax | 0-85 days after dosing
  Cmax
Pharmacokinetic parameters of ALIA-1758 in healthy subjects: T1/2 | 0-85 days after dosing
  elimination half-life (T1/2)
Pharmacokinetic parameters of ALIA-1758 in healthy subjects: AUC | 0-85 days after dosing
  Area Under Curve (AUC)
Pharmacokinetic parameters of ALIA-1758 in healthy subjects: Bioavailability | 0-85 days after dosing
  Bioavailability after SC administration (F)
Pharmacokinetic parameters of ALIA-1758 in healthy subjects: Clearance | 0-85 days after dosing
  Clearance (CL)
Pharmacokinetic parameters of ALIA-1758 in healthy subjects: Volume of distribution | 0-85 days after dosing
  Volume of distribution (Vz)

CONTACTS AND LOCATIONS:
Overall Officials: J. Michael Ryan, M.D., Study Director — AbbVie
Locations (1):
- Worldwide Clinical Trials Early Phase Services, LLC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No